CLINICAL TRIAL: NCT06618599
Title: Analgesic Effect of Mid-transverse Process to Pleura Block Combined With Erector Spinae Block Versus Paravertebral Plane Block in Thoracic Surgery for Lung Cancer Patients
Brief Title: Mid-transverse Process Combined With Erector Spinae Block Versus Paravertebral Plane Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sayed Mahmoud Abed, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: analgesia in thoracotomy
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Group 1: received ipsilateral Ultrasound guided midtransverse block and ipsilateral Ultrasound guided ESPB block Group 2: paravertebral block(PVB): Patients received ipsilateral Ultrasound guided paravertebral plane block .
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:midtransverse to pleura block combined with erector spinae block (Experimental): Patients received ipsilateral Ultrasound guided midtransverse block with injection of 20 ml bupivacaine 0.25% and ipsilateral Ultrasound guided ESPB block with injection of 20 ml bupivacaine 0.25%
  Interventions: Procedure: Mid-transverse process to pleura block combined with erector spinae block
- Group 2: paravertebral block (Experimental): Patients received ipsilateral Ultrasound guided paravertebral plane block with injection of 30 ml bupivacaine 0.25%.
  Interventions: Procedure: paravertebral block

INTERVENTIONS:
Procedure: Mid-transverse process to pleura block combined with erector spinae block — The probe will be placed vertically 3 cm lateral to the T5 spinous process and the transverse process will be identified. The needle will be introduced in an in-plane fashion until the tip lay deep in the erector spinae muscle. One milliliter of normal saline will be injected to confirm the correct needle tip position by visualizing the spread under the erector spinae muscle. 20 mL of 0.25% bupivacaine will be injected .The needle will be directed aiming for the midpoint between the transverse process and pleura from cephalad to caudad. One milliliter of normal saline will be given to confirm the position of the needle tip, then a total of 20 ml of 0.25% ropivacaine will be injected
  Arms: Group 1:midtransverse to pleura block combined with erector spinae block
Procedure: paravertebral block — the transducer will be positioned laterally 3 cm to the midline at T5 spinous process, defining the spinous process, pleura, transverse process, the paravertebral (PV) space, and superior costotransverse ligament. The trapezius, rhomboid major, and erector spinae muscles will be recognized as superficial to the hyperechoic transverse process shadow. However, when the rhomboid major muscle disappeared, this indicated that we will be at the 7th thoracic vertebra's level. Local infiltration using 2-3 mL of 2.0% lignocaine will be done. A spinal 22-gauge needle will be injected at the cephalic side of the transducer using an in-plane technique, and the needle directed towards the costotransverse ligament (CTL). The passage of the needle through the CTL will be associated with a pop, informing that the superior costotransverse ligament will be passed. Following a 3 mL testing dose of normal saline containing epinephrine (1:200,000), 30 mL bupivacaine 0.25% injected.
  Arms: Group 2: paravertebral block

SUMMARY:
This study aims to compare efficacy of Mid-transverse process to pleura block combined with erector spinae block versus paravertebral plane block in cancer patients undergoing thoracotomy surgeries.

DETAILED DESCRIPTION:
Thoracic paravertebral block (TPVB) application has also been used in recent years due to the lower incidence of side effects. The erector spinae plane block (ESPB)has been used as a part of multimodal analgesia in recent years. In ESPB is aimed to treat the postoperative pain of the thoracoabdominal region by injecting a local anesthetic into the interfacial area under the erector spinae muscle . ESPB creates an effect that covers the posterior and lateral thorax by affecting the dorsal rami and branches of the spinal nerves . Midtransverse process to pleura (MTP) block is less invasive as the position of the needle in this block is midway between the transverse process' posterior border and the pleura. Due to fenestrations present in the superior costotransverse ligament (SCTL), the drug reaches the paravertebral space

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patients for thoracotomy surgeries.
* Physical status American Society of Anesthesiologists (ASA )II, III.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2

Exclusion Criteria:

* Patient refusal
* physical status ASA IV,
* Age <18 years or >65 years
* BMI < 20 kg/m2 and >35 kg/m2
* Known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).
* History of psychological disorders and/or chronic pain.
* Contraindication to regional anesthesia e.g., local sepsis, pre- existing peripheral neuropathies, and coagulopathy.
* Severe respiratory, cardiac, hepatic or renal disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue score changes during rest and cough for the three groups. | for 24 hours postoperative
  the score of visual analogue score, with minimum score of 0 and maximum of 10, with higher scores meaning more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: sayed M Abed, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
starting from march 2025
Supporting Information: Study Protocol
Time Frame: basal
Access Criteria: web

REFERENCES:
- [Background] Zengin M, Alagoz A. Comparison of Thoracic Epidural Analgesia and Thoracic Paravertebral Block Applications in the Treatment of Acute Pain After Thoracotomy in Geriatric Patients. Cureus. 2021 Oct 22;13(10):e18982. doi: 10.7759/cureus.18982. eCollection 2021 Oct. PMID 34820237
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Liu L, Ni XX, Zhang LW, Zhao K, Xie H, Zhu J. Effects of ultrasound-guided erector spinae plane block on postoperative analgesia and plasma cytokine levels after uniportal VATS: a prospective randomized controlled trial. J Anesth. 2021 Feb;35(1):3-9. doi: 10.1007/s00540-020-02848-x. Epub 2020 Sep 4. PMID 32886200
- See also: https://jag.journalagent.com/scie/pdfs/SCIE-68926-RESEARCH_ARTICLE-BUKAGIKIRAN.pdf — https://jag.journalagent.com/scie/pdfs/SCIE-68926-RESEARCH_ARTICLE-BUKAGIKIRAN.pdf